CLINICAL TRIAL: NCT01705392
Title: A Randomized Phase II Trial Comparing Bevacizumab Monotherapy With Dacarbazine (DTIC) in Treatment of Malignant Melanoma, Focusing on Angiogenic Markers and Prevention of Hypertension.
Brief Title: Bevacizumab vs Dacarbazine in Metastatic Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of financing of the study drug. Not sufficient financial support.
Sponsor: Haukeland University Hospital (Other)
Collaborators: The Norwegian Melanoma Group (Unknown); Norwegian Cancer Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012/910
Record Dates: First submitted 2012-10-08; First posted 2012-10-12 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Metastatic Malignant Melanoma; Unresectable Malignant Melanoma
MeSH Terms: conditions — Melanoma | interventions — Bevacizumab; Propranolol; Enalapril; Enalaprilat; Dacarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Bevacizumab plus propranolol (Experimental): Bevacizumab 10mg/kg q2w plus propranolol 80 mg x 1
  Interventions: Drug: Bevacizumab; Drug: Propranolol
- Bevacizumab plus enalapril (Experimental): Bevacizumab 10mg/kg q2w plus enalapril 5 mg x 1
  Interventions: Drug: Bevacizumab; Drug: Enalapril
- Dacarbazine (Active Comparator): Dacarbazine 1000mg/m2 q3w
  Interventions: Drug: Dacarbazine

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab 10 mg/kg q3w
  Other Names: Avastin
  Arms: Bevacizumab plus enalapril; Bevacizumab plus propranolol
Drug: Propranolol — Propranolol 80 mg x 1
  Other Names: Inderal; Inderal retard
  Arms: Bevacizumab plus propranolol
Drug: Enalapril — Enalapril 5 mg x 1
  Other Names: Renitec; Vasotec
  Arms: Bevacizumab plus enalapril
Drug: Dacarbazine — dacarbazine 1000 mg/m2 q3w
  Other Names: DTIC
  Arms: Dacarbazine

SUMMARY:
The purpose of this study is to compare efficacy of bevacizumab monotherapy with standard chemotherapy (DTIC) in patients with metastatic malignant melanoma. In addition, we want to evaluate the predictive value of a set biomarkers associated with vascular endothelial growth factor (VEGF) dependent angiogenesis. Also, we aim to identify mechanisms causing acquired resistance to treatment with bevacizumab and escape mechanisms caused by other angiogenic growth factors than VEGF. Finally, we want to analyze safety and influence on outcome variables by primary prevention of bevacizumab induced hypertension by low dose beta blockers in comparison with an ACE inhibitor.

ELIGIBILITY:
Inclusion Criteria:

* Previously treated or untreated, histologically confirmed, metastatic and unresectable melanoma with progressive disease
* Both BRAF wild type patients as well as BRAF mutated patients are allowed. For BRAF mutated patients, BRAF targeting agents should be considered in first line if otherwise indicated and no contraindications exist.
* WHO performance status 0-1
* Age >18 years,
* Known BRAF mutation
* Able to undergo outpatient treatment
* Patients must have clinically and/or radiographically documented measurable disease according to RECIST.
* All radiology studies must be performed within 28 days prior to registration (35 days if negative).
* At least 4 weeks since adjuvant interferon alpha
* At least 4 weeks since 1st line treatment in case of metastasis
* Major surgical procedure or significant traumatic injury > 28 days prior to study treatment start. Biopsy or fine needle aspiration > 2 days prior to study treatment start. Central venous line placement must be inserted at least 2 days prior to treatment start.
* Only patients with irradiated and asymptomatic brain metastases and off dexamethasone are allowed.
* Hematology: absolute granulocytes > 1.0 x 109/L
* Platelets > 100 x 109/L
* Bilirubin < 1.5 x upper normal limit
* Serum creatinine < 1.5 x upper normal limits
* LDH < 1.5 x upper normal limit
* INR < 1.5
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial
* Before patient registration/randomization, written informed consent must be given according to national and local regulations.

Exclusion Criteria:

* No previous DTIC
* No previous anti-VEGF targeted therapies
* No pregnant or lactating patients can be included
* No clinical evidence of coagulopathy
* No unstable angina pectoris
* No AV-block II or III without pacemaker
* No severe congestive heart failure
* No untreated phaeochromocytoma
* No severe bradycardia
* No severe hypotension
* No severe impairment of peripheral arterial circulation
* No uncontrolled cardiac arrhythmia
* No severe asthma or COPD
* No uncontrolled diabetes mellitus
* No Angioneurotic edema
* No severe Aortic valve stenosis
* No severe hypertrophic cardiomyopathy
* No severe renal dysfunction
* No patients on beta blockers/ ACE inhibitors by inclusion unable/unwilling to discontinue beta blockers/ ACE inhibitors and convert to other classes of antihypertensive drugs
* No full-dose oral coumarin-derived anticoagulants (INR>1.5) or heparin, thrombolytic agents, or chronic, daily treatment with aspirin (>325 mg/day).
* No uncontrolled hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2017-02-20 (Actual); Study Completion 2017-02-20 (Actual)

PRIMARY OUTCOMES:
Progression free survival | Average of 6 months
  Participants will be followed for the duration of the treatment and as long as they do not progress, an expected average of 6 months

SECONDARY OUTCOMES:
Response Rates according to RECIST | Average 6 months
  Participants will be followed for the duration of the treatment with CT scans for response evaluation every 2 months for an expected average of 6 months.
Disease control rate at 6 months | 6 months
  Number of patient with complete response, partial response or stable disease at 6 months
Prevention of hypertension by beta blockers or ACE-inhibitors | Average of 6 months
  Safety and influence on outcome variables by primary prevention of bevacizumab induced hypertension, by low dose beta blockers (propranolol 80 mg x 1), in comparison with an ACE inhibitor (enalapril 5 mg x 1). Patients will be monitored as during active treatment with anti hypertensive drugs and bevacizumab for an average of 6 months.
Overall survival | Average og 12 months
  Participants will be followed until death for overall survival data, an expected average of 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Oddbjorn Straume, MD PhD, Principal Investigator — Department of Oncology, Haukeland University Hospital, Bergen, Norway; Olav Mella, MD PhD, Study Director — Department of Oncology, Haukeland University Hospital, Bergen, Norway
Locations (1):
- Haukeland University Hospital, Bergen, Norway